CLINICAL TRIAL: NCT03896074
Title: Phase II Randomized Trial Comparing Atezolizumab Versus Atezolizumab Plus Bevacizumab as First-line Treatment in PD-L1+ Advanced Metastatic Non-small-cell Lung Cancer Patients
Brief Title: Atezolizumab Versus Atezolizumab Plus Bevacizumab as First Line in NSCLC Patients (BEAT)
Acronym: BEAT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Ricerca Traslazionale (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FoRT 05- BEAT
Record Dates: First submitted 2019-03-04; First posted 2019-03-29 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Non-small-cell Lung Cancer Patients
MeSH Terms: interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atezolizumab (Experimental): Patients allocated to Arm A will be treated with atezolizumab administered intravenously at 1200 mg every 3 weeks given until disease progression, toxicity or patient refusal
  Interventions: Drug: Atezolizumab
- Atezolizumab plus bevacizumab (Experimental): Patients in the Arm B will receive atezolizumab administered intravenously at 1200 mg every 3 weeks plus bevacizumab intravenously at 15 mg/kg every 3 weeks given until disease progression, toxicity or patient refusal
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab administered intravenously at 1200 mg every 3 weeks
Drug: Bevacizumab — Bevacizumab intravenously at 15 mg/kg every 3 weeks
  Arms: Atezolizumab plus bevacizumab

SUMMARY:
phase II controlled randomized study comparing atezolizumab as single agent to the combination of atezolizumab and bevacizumab in patients with chemonaive metastatic NSCLC with PD-L1 expression. All NSCLC patients with tumor tissue available for biomarker assessment and candidate for first-line therapy are considered eligible for the study. After evaluation of all inclusion and exclusion criteria and after informed consent signature all eligible patients will be randomized to atezolizumab (Arm A) or to the combination of atezolizumab and bevacizumab (Arm B). Disease assessment will be performed every 6 weeks.

DETAILED DESCRIPTION:
This is a phase II controlled randomized study comparing atezolizumab as single agent to the combination of atezolizumab and bevacizumab in patients with chemonaive metastatic NSCLC with PD-L1 expression.

A total of maximum of 206 patients will be enrolled in the study. Patients will be treated with atezolizumab (1200 mg) every 3 weeks (6-week cycles) or the combination of atezolizumab (1200 mg) every 3 weeks (6-week cycles) plus bevacizumab (15 mg/kg) every 3 weeks until disease progression, unacceptable toxicity or patient refusal. Disease evaluation, along with various assessments, will be made every 3 weeks and every 6 weeks and follow-up every 3 months. Toxicities will be evaluated throughout the study period. A follow-up of 12 months is planned for each patient from the end of treatment .The study will be performed in approximately 20 centers across Italy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of stage IV non-squamous NSCLC with no evidence of EGFR sensitizing mutations or ALK or ROS1 rearrangements.
2. Availability of tumor tissue.
3. Evidence of PD-L1 expression evaluated with immunohistochemistry (≥1%).
4. No previous chemotherapy. Patients who have received prior neo-adjuvant, adjuvant chemotherapy, radiotherapy or chemoradiotherapy with curative intent for non-metastatic disease must have experienced a treatment-free interval of at least 6 months from randomization since the last dose of chemotherapy and/or radiotherapy.
5. ECOG performance status 0-1.
6. Life expectancy > 3 months
7. Age ≥18 years.
8. Measurable disease, as defined by RECIST v1.1.
9. Adequate hematologic and organ function, defined by the following laboratory results obtained within 28 days prior to randomization:

   * ANC ≥ 1500 cells/μL without granulocyte colony-stimulating factor support
   * Platelet count ≥ 100,000/μL without transfusion
   * Hemoglobin ≥ 9.0 g/dL Patients may be transfused to meet this criterion
   * AST, ALT, and alkaline phosphatase ≤ 2.5 × ULN, with the following exceptions:
   * Patients with documented liver metastases: AST and/or ALT ≤ 5 × ULN
   * Patients with documented liver or bone metastases: alkaline phosphatase ≤ 5 × ULN.
   * Serum bilirubin ≤ 1.25 × ULN
   * Patients with known Gilbert disease who have serum bilirubin level ≤ 3 mg/dL may be enrolled
   * Calculated creatinine clearance (CRCL) ≥ 45 mL/min or calculated CRCL must be ≥ 60 mL/min
10. Patient compliance to trial procedures.
11. Written informed consent.

Exclusion Criteria:

1. No tumor tissue available.
2. PD-L1 expression < 1 % or PD-L1 expression unknown or not assessable
3. Patient positive for EGFR mutations or ALK or ROS1 rearrangements.
4. Patients with squamous histology or with specific contraindication to bevacizumab therapy.
5. Previous chemotherapy. Adjuvant or neoadjuvant chemotherapy is considered a line of therapy if completed less than 6 months before evidence of disease relapse.
6. Concomitant radiotherapy or chemotherapy.
7. Previous therapy with any checkpoint inhibitor.
8. Pregnancy or lactating women who are pregnant, lactating, or intending to become pregnant during the study.
9. Symptomatic brain metastases; asymptomatic brain metastases are accepted if no steroid therapy is required and if pretreated.
10. Spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for > 2 weeks prior to randomization.
11. Leptomeningeal disease.
12. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently). Patients with indwelling catheters (e.g., PleurX) are allowed.
13. Uncontrolled or symptomatic hypercalcemia (> 1.5 mmol/L ionized calcium or Ca > 12 mg/dL or corrected serum calcium >ULN). Patients who are receiving denosumab prior to randomization must be willing and eligible to receive a bisphosphonate instead while on study.
14. Malignancies other than NSCLC within 5 years prior to randomization, with the exception of those with a negligible risk of metastasis or death (e.g., expected 5-year OS> 90%) treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, ductal carcinoma in situ treated surgically with curative intent)
15. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
16. Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the Atezolizumab formulation
17. History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, psoriatic arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. Patients with: 1) history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone, 2) controlled Type I diabetes mellitus who are receiving a stable dose of insulin regimen and 3) eczema, psoriasis, lichen simplex chronicus of vitiligo with dermatologic manifestations only in less than 10% of body surface area, well controlled at baseline and only requiring low potency topical steroids are eligible for this study.
18. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
19. Positive test for HIV
20. Patients with active hepatitis B (chronic or acute; defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C. Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as the presence of hepatitis B core antibody [HBc Ab] and absence of HBsAg) are eligible. HBV DNA must be obtained in these patients prior to randomization. Patients positive for hepatitis C virus (HCV) antibody are eligible only if PCR is negative for HCV RNA.
21. Active tuberculosis
22. Severe infections within 4 weeks prior to randomization, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia received therapeutic oral or IV antibiotics within 2 weeks prior to randomization. Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or to prevent chronic obstructive pulmonary disease exacerbation) are eligible.
23. Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within 3 months prior to randomization, unstable arrhythmias, or unstable angina. Patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or left ventricular ejection fraction < 50% must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate.
24. Major surgical procedure other than for diagnosis within 28 days prior to randomization or anticipation of need for a major surgical procedure during the course of the study
25. Prior allogeneic bone marrow transplantation or solid organ transplant
26. Administration of a live, attenuated vaccine within 4 weeks before randomization or anticipation that such a live attenuated vaccine will be required during the study
27. Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
28. Any approved anti-cancer therapy, including chemotherapy, or hormonal therapy within 3 weeks prior to initiation of study treatment; the following exceptions are allowed: Hormone-replacement therapy or oral contraceptives, TKIs approved for treatment of NSCLC discontinued > 7 days prior to randomization; the baseline scan must be obtained after discontinuation of prior TKIs.
29. Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 28 days prior to randomization
30. Prior treatment with CD137 agonists or immune checkpoint blockade therapies, anti-PD-1, and anti-PD-L1 therapeutic antibodies. Patients who have had prior anti-CTLA-4 treatment may be enrolled, provided the following requirements are met: Minimum of 6 weeks from the last dose of anti-CTLA-4; No history of severe immune-mediated adverse effects from anti-CTLA-4 (NCI CTCAE Grade 3 and 4)
31. Treatment with systemic immunostimulatory agents (including but not limited to IFNs, IL-2) within 6 weeks or five half-lives of the drug, wichever is shorter, prior to randomization. Prior treatment with cancer vaccines is allowed.
32. Treatment with systemic immunosuppressive medications (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to randomization.
33. Patients who have received acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled in the study after discussion with and approval by the Medical Monitor.
34. Patients with history of allergic reaction to IV contrast requiring steroid pre-treatment should have baseline and subsequent tumor assessments done by MRI. The use of inhaled corticosteroids for chronic obstructive pulmonary disease, mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension, and low-dose supplemental corticosteroids for adrenocortical insufficiency are allowed.
35. Inadequately controlled hypertension (defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg) Anti-hypertensive therapy to achieve these parameters is allowable.
36. Prior history of hypertensive crisis or hypertensive encephalopathy
37. Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recentperipheral arterial thrombosis) within 6 months prior to randomization
38. History of hemoptysis (≥ one-half teaspoon of bright red blood per episode) within 1 month prior to randomization; Evidence of bleeding diathesis or coagulopathy (in the absence of therapeutic anticoagulation).
39. Current or recent (within 10 days of randomization) use of aspirin (> 325 mg/day) or treatment with dipyramidole, ticlopidine, clopidogrel, and clostazol
40. Current use of full-dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic purposes that has not been stable for > 2 weeks prior to randomization. The use of full-dose oral or parenteral anticoagulants is permitted as long as the INR or aPTT is within therapeutic limits (according to the medical standard of the enrolling institution) and the patient has been on a stable dose of anticoagulants for at least 2 weeks prior to randomization.
41. Prophylactic anticoagulation for the patency of venous access devices is allowed, provided the activity of the agent results in an INR< 1.5 ×ULN and aPTT is within normal limits within 14 days prior to randomization.
42. Prophylactic use of low-molecular-weight heparin (i.e., enoxaparin 40 mg/day) is permitted.
43. Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to the first dose of bevacizumab
44. History of abdominal or tracheosphageal fistula or gastrointestinal perforation within 6 months prior to randomization; Clinical signs of gastrointestinal obstruction or requirement for routine parenteral hydration, parenteral nutrition, or tube feeding; Evidence of abdominal free air not explained by paracentesis or recent surgical procedure.
45. Serious, non-healing wound, active ulcer, or untreated bone fracture
46. Proteinuria, as demonstrated by urine dipstick or > 1.0 g of protein in a 24-hour urine collection. All patients with ≥ 2+ protein on dipstick urinalysis at baseline must undergo a 24-hour urine collection and must demonstrate ≤ 1 g of protein in 24 hours.
47. Known sensitivity to any component of bevacizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2020-03-02 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | 18 months
  Overall Survival (OS) rate at 18 months in patients treated with atezolizumab alone versus atezolizumab-bevacizumab combination

SECONDARY OUTCOMES:
Response rate (complete + partial responses) | Up to 24 months
  Response rate will be evaluated by investigators according to RECIST criteria version 1.1. Partial and complete responses will be confirmed following RECIST criteria 1.1.
Progression-free survival | Up to 24 months
  Progression free survival (PFS) will be calculated from the date of randomization to the first documented evidence of progressive disease or death due to any cause (whichever occurs first).
Overall survival according to presence of bone and/ or hepatic metastases | Up to 24 months
  Overall response rate (ORR) is defined as the number of subjects with a best overall response (BOR) of CR or PR divided by the number of randomized subjects for each treatment group.

CONTACTS AND LOCATIONS:
Locations (33):
- Italy (33):
  - Ospedale Degli Infermi Di Biella, Ponderano, BI
  - Asst Di Lecco, Lecco, CM
  - A.O.U. Policlinico - Vittorio Emanuele- Presidio Ospedaliero Gaspare Rodolico, Catania, CT
  - Ospedale Della Misericordia, Grosseto, GR
  - Presidio Ospedaliero Unico Av3 - Ospedale Generale Provinciale - Macerata, Macerata, MC
  - Fondazione IRCCS - San Gerardo del Tintori, Monza, MILANO
  - Azienda Ospedaliero-Universitaria Di Modena, Modena, MO
  - AZIENDA USL DI PIACENZA-Ospedale Guglielmo da Saliceto, Piacenza, PC
  - C.R.O.B. - I.R.C.C.S., Rionero in Vulture, PZ
  - AUSL della Romagna, Ravenna, RA
  - OSPEDALE SAN PAOLO - ASL Roma 4, Civitavecchia, RM
  - Fondazione PTV - POLICLINICO TOR VERGATA, Roma, RM
  - Azienda Ospedaliera S.Giovanni Addolorata, Roma, RM
  - Azienda Ospedaliera San Camillo-Forlanini, Roma, Roma
  - P.O. Umberto I, Syracuse, SR
  - Ospedale S.G. Moscati, Statte, TA
  - AUSL di Teramo - Ospedale "Giuseppe Mazzini", Teramo, TE
  - AOU Ospedali Riuniti "Umberto I- G.M.Lancisi-G.Salesi", Ancona
  - IRCCS Oncologico Istituto Tumori "Giovanni Paolo II", Bari
  - P.O. Antonio Perrino, Brindisi
  - A.O. Per l' emergenza Cannizzaro, Catania
  - Irccs S.R.L. Irst, Meldola
  - AO Papardo, Messina
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera Dei Colli V.Monaldi, Napoli
  - Istituto Nazionale Tumori di Napoli IRCCS Pascale, Napoli
  - Ospedale Sacro Cuore- Don Calabria, Negrar
  - AOU S. Luigi Orbassano, Orbassano
  - IRCCS ISTITUTO Oncologico Veneto, Padua
  - Arcispedale Santa Maria Nuova, Reggio Emilia
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - ASST Sette Laghi, Varese
  - AUOI di Verona- Borgo Trento, Verona